CLINICAL TRIAL: NCT07322757
Title: Outcomes-Based Health Program for Improving Care and Outcomes in Patients With Type 2 Diabetes: A Real-World Implementation Study in Primary Care
Brief Title: Outcomes-Based Health Program for Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Finnish Diabetes Association (Other); University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Sonja Soininen, Physician in Chief, Teaching clinic Osmo, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5103906
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; High-risk type 2 diabetes patients; Digital lifestyle intervention; PROM; PAID
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital intervention arm (Experimental): Digital interventions: BitHabit application and optionally Onnikka application
  Interventions: Other: BitHabit digital application for behavioral lifestyle changes; Other: Onnikka weight management digital application
- Control group (No Intervention): Control group receives same enhancement in treatment plan, but no digital interventions

INTERVENTIONS:
Other: BitHabit digital application for behavioral lifestyle changes — BitHabit digital application for behavioral lifestyle changes
  Arms: Digital intervention arm
Other: Onnikka weight management digital application — Onnikka weight management digital application
  Arms: Digital intervention arm

SUMMARY:
Type 2 diabetes is a growing health concern worldwide, influenced by genetic factors, overweight, metabolic syndrome, and insufficient physical activity. Good treatment and glycemic control can reduce or delay diabetes-related complications, which account for a significant and increasing share of healthcare costs in Finland. Much of this cost growth is due to complications resulting from inadequate diabetes care. Secondary prevention programs can therefore provide both health and economic benefits. Lifestyle interventions are one way to improve type 2 diabetes care and reduce complications.

This study aims to evaluate the impact of a digital lifestyle intervention combined with optimized care on treatment and outcomes among adults with type 2 diabetes at high risk for complications.

The intervention includes access to the BitHabit "Small Actions" application, which supports healthy lifestyle changes, and for participants with a body mass index (BMI) over 30, the Onnikka weight management application. The study will be conducted in North Savo, Finland, using a case-control design. Approximately 120 participants will receive the intervention and 50-100 will serve as controls. All participants will have their care plans reviewed and updated according to the Finnish Current Care Guidelines for Type 2 Diabetes. Control group participants will receive standard care, while the intervention group will receive standard care plus the digital tools. The study also includes the validation of the PAID (Problem Areas in Diabetes) questionnaire for use in Finland and in the Finnish language.

The study duration for each participant is 12 months. Data will be collected through physiological measurements, laboratory tests, questionnaires, and app usage logs. Measurements and questionnaires will be conducted at baseline and after 12 months. The analyses will describe the phenomenon, its prevalence, and associations between variables, as well as potential dependencies.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed
* At least one of the following:

  1. diagnosed coronary artery disease,
  2. diagnosed periferal artery disease,
  3. diagnosed heart failure,
  4. diagnosed diabetic renal disease (GFR <60 OR uACR ≥ 3 for at least three months),
  5. diagnosed diabetic retinopathy,
  6. previous stroke,
  7. diagnosed atrial fibrillation or atrial flutter,
  8. age ≥ 55 years and at least two of the following conditions:

     1. smoker
     2. uses antihypertensive medication or systolic blood pressure >140 mmHg or diastolic blood pressure > 80 mmHg,
     3. uses lipid lowering medication or LDL-cholesterol > 2.6 or
     4. BMI > 25

Exclusion Criteria:

* eGFR < 30
* uACR > 200
* BMI > 50
* heart ejection fraction EF < 30
* active cancer or less than five years from cancer treatment at enrollment
* blindness in both eyes
* severe psychotic depression
* inability to utilize digital applications

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in weight at 12 months | From enrollment to the end of follow-up at 12 months
  Change from baseline in weight at 12 months. Weight measurement is taken by study nurse both at baseline and at the end of the study.
Change from baseline in BMI at 12 months | From enrollment to the end of follow-up at 12 months
  Change from baseline in BMI at 12 months. Weight and height measurement are taken by study nurse both at baseline and at the end of the study.
Change from baseline in waist circumference at 12 months | From enrollment to the end of follow-up at 12 months
  Change from baseline in waist circumference at 12 months. Waist circumference is taken by study nurse both at baseline and at the end of the study.
Change from baseline in Body Roundness Index at 12 months | From enrollment to the end of follow-up at 12 months
  Change from baseline in Body Roundness Index at 12 months. Weight, height, waist and hip circumference are taken by study nurse both at baseline and at the end of the study.
Change from baseline in HbA1c at 12 months | From enrollment to the end of follow-up at 12 months
  Change from baseline in HbA1c at 12 months. HbA1c is a laboratory measurement describing glucose levels, taken both at baseline and at the end of the study.
Change from baseline in serum lipid levels at 12 months | From enrollment to the end of follow-up at 12 months
  Change from baseline in serum lipid levels at 12 months. LDL, HDL and triglycerides are laboratory measurements taken both at baseline and at the end of the study.
Change from baseline in smoking status at 12 months | From enrollment to the end of follow-up at 12 months
  Change from baseline in smoking status at 12 months. Smoking status is surveyed both at baseline and at the end of the study.
Change from baseline in physical activity at 12 months | From enrollment to the end of follow-up at 12 months
  Change from baseline in physical activity at 12 months. Physical activity is surveyed both at baseline and at the end of the study.
Change from baseline in dietary habits at 12 months | From enrollment to the end of follow-up at 12 months
  Change from baseline in dietary habits at 12 months. Dietary habits are surveyed both at baseline and at the end of the study.
Change from baseline in blood pressure at 12 months | From enrollment to the end of follow-up at 12 months
  Change from baseline in blood pressure at 12 months. Blood pressure measurement is taken by study nurse via Riva Rocci method both at baseline and at the end of the study.
Self-reported changes from baseline in qualty of life measured by EQ-5D-5L at 12 months | From enrollment to the end of follow-up at 12 months
  EQ-5D-5L is a standard health questionnaire assessing quality of life across five dimensios: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. EQ-5D-5L questionnaire is filled electronically at baseline and at the end of the study.
Change from baseline in Problem Areas in Diabetes (PAID) scale at 12 months | From enrollment to the end of follow-up at 12 months
  PAID scale identifies emotional distress in diabetes, covering issues like worrying complications, goal setting, food, treatment, and social support, common problems including fear, anger, feeling overwhelmed and guilt.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Soininen, MD, PhD, Principal Investigator — Wellbeing Services County of North Savo, Kuopio, Finland
Locations (1):
- Wellbeing services county of North Savo, Nursing and Physician Services, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No
Study permission does not allow sharing individual participant data.